CLINICAL TRIAL: NCT05283525
Title: Efficacy Of Trimrox On Body Composition, Body Weight, And Anthropometric Parameters In 100 Healthy Male And Female Volunteers
Brief Title: Efficacy Of Trimrox On Body Recomposition And Weight Management (TRCAP21)
Acronym: VNI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Victory Nutrition International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: VNI-TRIMROX-2022
Record Dates: First submitted 2022-01-10; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-02

CONDITIONS: Body Weight Changes
Keywords: TrimRox (TRCAP21); 90-Day Investigation; 100 Subjects; Body Weight, Height, Body Mass Index (BMI); Blood Pressure; Anthropometric Measurement; Body Composition; Oxygen Saturation; Adverse Event Monitoring
MeSH Terms: conditions — Body Weight Changes; Body Weight | interventions — Oxygen Saturation; Sleep; Health Status

STUDY DESIGN:
Intervention Model Description: A Longitudinal Study To Determine The Efficacy of Trimrox Efficacy On Body Recomposition And Weight Management In Human Volunteers
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind placebo-controlled study. An independent body will randomize the study subjects and determine the placebo- and treatment group subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Group #1 (6.75 gms Once-A-Day) (Placebo Comparator): Placebo Group #1 (1 Dose; 6.75 gms per day): A total of 25 subjects will be given 1 placebo sachet; To be taken one in the morning in an empty stomach over a period of 90 consecutive days
  Interventions: Dietary Supplement: Anthropometric Measurement of the Chest, Upper Arm/Bicep, Hips, Thighs and Waist/ Belly in Inches; Dietary Supplement: Oxygen Saturation; Dietary Supplement: Total Blood Chemistry; Dietary Supplement: Adverse Event Monitoring; Dietary Supplement: Body Weight Monitoring; Dietary Supplement: Physical well-being including mood, energy, satiety level. sugar cravings, sleep, and overall health
- Placebo Group #2 (6.75 gms Twice-A-Day) (Placebo Comparator): Placebo Group #2 (2 Doses; 13.5 gms in two divided doses per day): A total of 25 subjects will be given 2 placebo sachets; To be taken one in the morning in an empty stomach and the other in the afternoon in an empty stomach over a period of 90 consecutive days
  Interventions: Dietary Supplement: Anthropometric Measurement of the Chest, Upper Arm/Bicep, Hips, Thighs and Waist/ Belly in Inches; Dietary Supplement: Oxygen Saturation; Dietary Supplement: Total Blood Chemistry; Dietary Supplement: Adverse Event Monitoring; Dietary Supplement: Body Weight Monitoring; Dietary Supplement: Physical well-being including mood, energy, satiety level. sugar cravings, sleep, and overall health
- TRCAP21 Group #1 (6.75 gms Once-A-Day) (Active Comparator): TRCAP21 Group #1 (1 Dose; 6.75 gms per day): A total of 25 subjects will be given 1 TRCAP21 sachet; To be taken one in the morning in an empty stomach over a period of 90 consecutive days
  Interventions: Dietary Supplement: Anthropometric Measurement of the Chest, Upper Arm/Bicep, Hips, Thighs and Waist/ Belly in Inches; Dietary Supplement: Oxygen Saturation; Dietary Supplement: Total Blood Chemistry; Dietary Supplement: Adverse Event Monitoring; Dietary Supplement: Body Weight Monitoring; Dietary Supplement: Physical well-being including mood, energy, satiety level. sugar cravings, sleep, and overall health
- TRCAP21 Group #2 (6.75 gms Twice-A-Day) (Active Comparator): TRCAP21 Group #2 (2 Doses; 13.5 gms in two divided doses per day): A total of 25 subjects will be given 2 TRCAP21 sachets; To be taken one in the morning in empty stomach and the other in the afternoon in an empty stomach over a period of 90 consecutive days
  Interventions: Dietary Supplement: Anthropometric Measurement of the Chest, Upper Arm/Bicep, Hips, Thighs and Waist/ Belly in Inches; Dietary Supplement: Oxygen Saturation; Dietary Supplement: Total Blood Chemistry; Dietary Supplement: Adverse Event Monitoring; Dietary Supplement: Body Weight Monitoring; Dietary Supplement: Physical well-being including mood, energy, satiety level. sugar cravings, sleep, and overall health

INTERVENTIONS:
Dietary Supplement: Anthropometric Measurement of the Chest, Upper Arm/Bicep, Hips, Thighs and Waist/ Belly in Inches — 0 - 90 Days of Treatment
  Other Names: Anthropometric Measurements
Dietary Supplement: Oxygen Saturation — 0 - 90 Days of Treatment
Dietary Supplement: Total Blood Chemistry — 0 and 90 Days of Treatment
Dietary Supplement: Adverse Event Monitoring — Adverse Event Monitoring Throughout the Study
Dietary Supplement: Body Weight Monitoring — 0 - 90 Days of Treatment
  Other Names: Adverse Event Monitoring in All Groups
Dietary Supplement: Physical well-being including mood, energy, satiety level. sugar cravings, sleep, and overall health — 0 - 90 Days of Treatment
  Other Names: Physical well-being

SUMMARY:
Protocol Number: VNI/121/TrimRox:

A unique stimulant- and sugar-free TRCAP21 Prodosomed® nutraceutical formulation, TrimROXTM, has been developed in a cGMP and NSF-certified manufacturing facility that is CFR-111 A compliant as well as having a BRC A rating, ensuring compliance with the Global Food Safety Initiative (GFSI). The investigators developed a stimulant- and sugar-free TRCAP21 Prodosomed® nutraceutical technology that effectively addresses directly and indirectly all the contributing factors. The investigators will conduct a 90-day study investigation in 100 study participants to assess the efficacy of TRCAP21 on diverse anthropometric aspects including chest, upper arms, waist/belly, hips and thighs, body weight, height, body mass index (BMI), and overall health and well-being.

DETAILED DESCRIPTION:
CDC reports that in the USA, the prevalence of obesity was 40% in adults between 20 and 39 years, 44.8% in adults between 40 and 59 years, and 42.8% in people 60 years and older. Furthermore, the CDC emphasized that 49.6% of non-Hispanic Black adults exhibited the highest age-adjusted prevalence of obesity, which is followed by the occurrence of 44.8% in Hispanic adults, 42.2% in non-Hispanic White adults, and 17.4% in non-Hispanic Asian adults. Obesity-related conditions include diverse cardiovascular diseases and dysfunctions, stroke, Type 2 Diabetes, and certain types of cancer that are some of the leading causes of preventable, premature death. The estimated annual medical cost of obesity in the United States was $147 billion in 2008 US dollars; the medical cost for people who have obesity was $1,429 higher than those of normal weight. Overall, the obesity epidemic is increasing at an alarming rate worldwide. Because of the alarming rise in the global obesity epidemic, the terminologies "weight loss" and "weight management" have become common descriptors, even in the medical and scientific communities. However, the correct scientific terminology should more accurately refer to express changes in body composition and size, especially in regard to a reduction in fat mass, rather than weight reduction alone. In fact, the investigators will demonstrate that focusing on "weight" as an appropriate measuring criterion constitutes a contradiction and a misconception to the natural sequence of metabolic events in the body recomposition process. Overall, the term 'weight loss' is an unreliable metric as it automatically places the primary focus on the heaviness of the body and does not provide a correct and accurate perspective for evaluating healthy changes in metabolism, body composition, or size. For example, losing a small amount of fat while increasing muscle density, strength, and performance could result in a small increase in weight, as muscle is heavier than fat. It is especially important to highlight that fat is the lightest of pertinent macro molecules in the human body, lighter than water, muscle mass, and bone. Moreover, fat is usually 'the last to go' in the body recomposition process, therefore, creating short-term expectations in weight loss is erroneous and maybe even fraudulent.

A more comprehensive and accurate approach therefore is to fundamentally restore healthy efficient aerobic metabolism, improving oxygen utilization and management that enables competent cellular waste removal. Adversarial factors to that objective involve nutrient deprivation (the most common factor employed by weight loss products and programs), the imposition of various types of stimulants inducing, via feedback, regulatory energy-conserving retaliation in the form of even greater survival insurance storage; triggering the "yo-yo" rebound weight regain. Moreover, conventional weight loss tactics seem to ignore the biological, genetic, and metabolic consequences that occur with aging. Diminishing hormonal potencies are crucially important considerations that need to be addressed in the obesity epidemic. Cellular oxygen deprivation-induced anaerobic pathologies exacerbate and amplify the effects of diminished hormone functionality and contribute to an increasingly sluggish metabolism with increased fat, glycogen, and water storage. This also increases the detrimental strain on the cardiovascular system, kidneys, GI tract, and microbiome to name a few. The objective is to restore optimal systemic aerobic metabolism using a novel TRCAP21 nutraceutical formulation that addresses multiple biological pathways in order to reduce survival panic, restore survival safety, and correct metabolic homeostasis.

ELIGIBILITY:
Inclusion Criteria

1. Agrees to sign written and audio-visual informed consent.
2. Fully understand the risks and benefits of the study
3. Male and Female Subjects (age: 30-70 Y)
4. Subjects are deemed to be acceptable for this study by their physician

Exclusion Criteria

1. Subjects who are unwilling or uncooperative subjects
2. Subjects were excluded who had impaired hepatic functions i,e., SGOT/SGPT >2.5 X
3. Subjects suffering from type 1 diabetes
4. Subjects suffering from type 2 diabetes or anyone else that has a blood glucose levels >180 mg/dl or HbA1c > 8.
5. Subjects who were suffering from coronary artery disease or high blood pressure >180/100
6. Subjects who were exhibiting abnormal hepatic or kidney functions (ALT or AST > 2 X greater than normal value); elevated creatinine, males > 125 μmol/L or 1.4mg/dl
7. Subjects who have cancer and are suffering from a malignancy.
8. Hypersensitivity to the investigational supplement
9. Subjects who had used any known weight management supplement for the last 2 months.
10. History of blood coagulation and bleeding (coagulopathies)
11. Incidence of high alcohol intake (more than 2 standard drinks/day).
12. Psychiatric disorder/disability provide signed informed consent.
13. Existing medical condition of the participant, which may be detrimental to the study and subject's overall well-being.

    __________________________________________________________________

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-23 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2024-01-09 (Estimated)

PRIMARY OUTCOMES:
Anthropometric Measurement of the Chest (in Inches) | 0 Day of Treatment
  Anthropometric Measurement of the Chest (in Inches)
Anthropometric Measurement of the Chest (in Inches) | 30 Day of Treatment
  Anthropometric Measurement of the Chest (in Inches)
Anthropometric Measurement of the Chest (in Inches) | 60 Day of Treatment
  Anthropometric Measurement of the Chest (in Inches)
Anthropometric Measurement of the Chest (in Inches) | 90 Days of Treatment
  Anthropometric Measurement of the Chest (in Inches)
Anthropometric Measurement of the Upper Arm/Bicep (in Inches) | 0 Day of Treatment
  Anthropometric Measurement of the Upper Arm/Bicep (in Inches)
Anthropometric Measurement of the Upper Arm/Bicep (in Inches) | 30 Days of Treatment
  Anthropometric Measurement of the Upper Arm/Bicep (in Inches)
Anthropometric Measurement of the Upper Arm/Bicep (in Inches) | 60 Days of Treatment
  Anthropometric Measurement of the Upper Arm/Bicep (in Inches)
Anthropometric Measurement of the Upper Arm/Bicep (in Inches) | 90 Days of Treatment
  Anthropometric Measurement of the Upper Arm/Bicep (in Inches)
Anthropometric Measurement of the Hip (in Inches) | 0 Day of Treatment
  Anthropometric Measurements of the Hip (in Inches)
Anthropometric Measurement of the Hip (in Inches) | 30 Days of Treatment
  Anthropometric Measurements of the Hip (in Inches)
Anthropometric Measurement of the Hip (in Inches) | 60 Days of Treatment
  Anthropometric Measurements of the Hip (in Inches)
Anthropometric Measurement of the Hip (in Inches) | 90 Days of Treatment
  Anthropometric Measurements of the Hip (in Inches)
Anthropometric Measurement of the Thighs (in Inches) | 0 Day of Treatment
  Anthropometric Measurement of the Thighs (in Inches)
Anthropometric Measurement of the Thighs (in Inches) | 30 Days of Treatment
  Anthropometric Measurement of the Thighs (in Inches)
Anthropometric Measurement of the Thighs (in Inches) | 60 Days of Treatment
  Anthropometric Measurement of the Thighs (in Inches)
Anthropometric Measurement of the Thighs (in Inches) | 90 Days of Treatment
  Anthropometric Measurement of the Thighs (in Inches)
Anthropometric Measurement of the Waist/Belly (in Inches) | 0 Day of Treatment
  Anthropometric Measurements of the Waist/Belly (in Inches)
Anthropometric Measurement of the Waist/Belly (in Inches) | 30 Days of Treatment
  Anthropometric Measurements of the Waist/Belly (in Inches)
Anthropometric Measurement of the Waist/Belly (in Inches) | 60 Days of Treatment
  Anthropometric Measurements of the Waist/Belly (in Inches)
Anthropometric Measurement of the Waist/Belly (in Inches) | 90 Days of Treatment
  Anthropometric Measurements of the Waist/Belly (in Inches)
Body Weight Measurement (in Kilograms) | 0 Day of Treatment
  Body Weight Measurements (in Kilograms)
Body Weight Measurement (in Kilograms) | 30 Days of Treatment
  Body Weight Measurements (in Kilograms)
Body Weight Measurement (in Kilograms) | 60 Days of Treatment
  Body Weight Measurements (in Kilograms)
Body Weight Measurement (in Kilograms) | 90 Days of Treatment
  Body Weight Measurements (in Kilograms)
Height Measurement (in Centimeters) | 0 Day of Treatment
  Height Measurement (in Centimeters)
Height Measurement (in Centimeters) | 30 Days of Treatment
  Height Measurement (in Centimeters)
Height Measurement (in Centimeters) | 60 Days of Treatment
  Height Measurement (in Centimeters)
Height Measurement (in Centimeters) | 90 Days of Treatment
  Height Measurement (in Centimeters)
BMI (body mass index) Measurement (in kg/m^2) | 0 Day of Treatment
  BMI (body mass index)(kg/m^2)
BMI (body mass index) Measurement (in kg/m^2) | 30 Days of Treatment
  BMI (body mass index)(kg/m^2)
BMI (body mass index) Measurement (in kg/m^2) | 60 Days of Treatment
  BMI (body mass index)(kg/m^2)
BMI (body mass index) Measurement (in kg/m^2) | 90 Days of Treatment
  BMI (body mass index)(kg/m^2)

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure Measurements (in mmHg) | 0 Day of Treatment
  Systolic and Diastolic Blood Pressure Measurements (mmHg)
Systolic and Diastolic Blood Pressure Measurements (in mmHg) | 30 Days of Treatment
  Systolic and Diastolic Blood Pressure Measurements (mmHg)
Systolic and Diastolic Blood Pressure Measurements (in mmHg) | 60 Days of Treatment
  Systolic and Diastolic Blood Pressure Measurements (mmHg)
Systolic and Diastolic Blood Pressure Measurements (in mmHg) | 90 Days of Treatment
  Systolic and Diastolic Blood Pressure Measurements (mmHg)
Pulse Rate Measurement (in beats per minute; bpm) | 0 Day of Treatment
  Pulse Rate (beats per minute; bpm)
Pulse Rate Measurement (in beats per minute; bpm) | 30 Days of Treatment
  Pulse Rate (beats per minute; bpm)
Pulse Rate Measurement (in beats per minute; bpm) | 60 Days of Treatment
  Pulse Rate (beats per minute; bpm)
Pulse Rate Measurement (in beats per minute; bpm) | 90 Days of Treatment
  Pulse Rate (beats per minute; bpm)
Saturation of Oxygen in Red Blood Cells (Pulse Ox Measurements; SpO2%) | 0 Day of Treatment
  Pulse Ox Measurement (SpO2%)
Saturation of Oxygen in Red Blood Cells (Pulse Ox Measurements; SpO2%) | 30 Days of Treatment
  Pulse Ox Measurement (SpO2%)
Saturation of Oxygen in Red Blood Cells (Pulse Ox Measurements; SpO2%) | 60 Days of Treatment
  Pulse Ox Measurement (SpO2%)
Saturation of Oxygen in Red Blood Cells (Pulse Ox Measurements; SpO2%) | 90 Days of Treatment
  Pulse Ox Measurement (SpO2%)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Bruce S. Morrison, Huntingdon Valley, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
YES
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Jan 23, 2022 to Jan 22, 2023
Access Criteria: www.vni.life
URL: http://www.vni.life